CLINICAL TRIAL: NCT02427581
Title: A Phase 1 Clinical Trial to Evaluate the Safety and Immunogenicity of a Personalized Synthetic Long Peptide Breast Cancer Vaccine Strategy in Patients With Persistent Triple-Negative Breast Cancer Following Neoadjuvant Chemotherapy
Brief Title: Safety and Immunogenicity of a Personalized Synthetic Long Peptide Breast Cancer Vaccine Strategy in Patients With Persistent Triple-Negative Breast Cancer Following Neoadjuvant Chemotherapy
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Drugs not available
Sponsor: Washington University School of Medicine (Other)
Collaborators: Susan G. Komen Breast Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201506113
Record Dates: First submitted 2015-04-22; First posted 2015-04-28 (Estimated); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Triple Negative Breast Cancer; Triple Negative Breast Neoplasms; Triple-Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — poly ICLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1 - personlized synthetic long peptide vaccine (Experimental): * Each subject will receive a single synthetic long peptide vaccine on Days 1, 4, 8, 15, 22, 50, and 78.
  * The first five injections must take place within +/- 1 day window and the remaining injections must take place within a +/- 2 week window.
  * The synthetic long vaccine is reconstituted in up to four pools (A, B, C, and D). At each vaccination time point, each of the up to four pools will be administered to one of the four limbs (A - Right Arm, B - Left Arm, C - Right Leg, and D - Left Leg) by subcutaneous (SC) injection. Alternative anatomical locations for patients who are status post complete axillary or inguinal lymph node dissection or other contraindications that prevent injections to a particular extremity are the left and right midriff, respectively. The same pool should be administered to the same limb across doses.
  Interventions: Biological: Personalized synthetic long peptide vaccine (Poly ICLC); Drug: Poly ICLC

INTERVENTIONS:
Biological: Personalized synthetic long peptide vaccine (Poly ICLC)
Drug: Poly ICLC
  Other Names: Hiltonol

SUMMARY:
The most important consideration in the design of this clinical trial is to ensure the safe translation of the personalized synthetic long peptide vaccine strategy. The Food and Drug Administration (FDA) dictates that initial studies of biologic therapies be performed in such a way that there is a balance between the potential risks and benefits in individual patients. Consistent with these recommendations, the investigators will target patients with triple-negative breast cancer who do not have a pathologic complete response after neoadjuvant chemotherapy. These patients typically have no gross evidence of disease following standard of care therapy (neoadjuvant chemotherapy, surgery and radiation therapy) but are at extremely high-risk for disease recurrence. Targeting this patient population provides a window-of-opportunity to design and manufacture the personalized cancer vaccines, maximizes the potential benefit from the vaccine as the regulatory networks associated with metastatic disease are not present, and balances risk in this patient population with extremely high risk for disease recurrence but no other treatment options.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of invasive breast cancer.
* ER and PR less than Allred score of 3 or less than 1% positive staining cells in the invasive component of the tumor
* HER2 negative by FISH or IHC staining 0 or 1+.
* Consented for genome sequencing and dbGAP-based data sharing and has provided or will provide germline and tumor DNA samples of adequate quality for sequencing. Fresh tissue is preferred (from biopsy at the time of port placement) but archival tissue is allowed.
* Clinical stage T2-T4c, any N, M0 primary tumor by AJCC 7th edition clinical staging prior to neoadjuvant chemotherapy, with residual invasive breast cancer after neoadjuvant therapy. If the patient has invasive cancer in the contralateral breast, she is not eligible for this study.
* At least 18 years of age.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Adequate organ and marrow function no more than 14 days prior to registration as defined below:

  * WBC ≥3,000/μL
  * absolute neutrophil count ≥1,500/μL
  * platelets ≥100,000/μL
  * total bilirubin ≤2.5 X institutional upper limit of normal
  * AST/ALT ≤2.5 X institutional upper limit of normal
  * creatinine ≤1.5 X institutional upper limit of normal
* Women of reproductive potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation.
* Able to understand and willing to sign an IRB-approved written informed consent document.

Exclusion Criteria:

* Evidence of progressive breast cancer within the last 30 days.
* Received chemotherapy, radiotherapy, or biologic therapy within the last 30 days (neoadjuvant chemotherapy excluded).
* Experiencing adverse events due to agents administered more than 30 days earlier.
* Receiving any other investigational agent(s) or has received an investigational agent within the last 30 days.
* Known metastatic disease.
* Invasive cancer in the contralateral breast.
* Known allergy, or history of serious adverse reaction to vaccines such as anaphylaxis, hives, or respiratory difficulty.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia (including sinus bradycardia), or psychiatric illness/social situation that would limit compliance with study requirements.
* Prior or currently active autoimmune disease requiring management with immunosuppression. This includes inflammatory bowel disease, ulcerative colitis, Crohn's disease, systemic vasculitis, scleroderma, psoriasis, multiple sclerosis, hemolytic anemia, immune-mediated thrombocytopenia, rheumatoid arthritis, systemic lupus erythematosus, Sjorgen's syndrome, sarcoidosis, or other rheumatologic disease or any other medical condition or use of medication (e.g., corticosteroids) which might make it difficult for the patient to complete the full course of treatments or to generate an immune response to vaccines. Asthma or chronic obstructive pulmonary disease that does not require daily systemic corticosteroids is acceptable. Any patients receiving steroids should be discussed with the PI to determine if eligible.
* Pregnant or breastfeeding. A negative serum pregnancy test is required no more than 7 days before study entry.
* The patient with a previous history of non-breast malignancy is eligible for this study only if the patient meets the following criteria for a cancer survivor. A cancer survivor is eligible provided the following criteria are met: (1) patient has undergone potentially curative therapy for all prior malignancies, (2) patients have been considered disease free for at least 1 year (with the exception of basal cell or squamous cell carcinoma of the skin or carcinoma-in-situ of the cervix).
* Patient must have no active major medical or psychosocial problems that could be complicated by study participation.
* Known HIV-positive status. These patients are ineligible because of the potential inability to generate an immune response to vaccines.
* Subjects with a strong likelihood of non-adherence such as difficulties in adhering to follow-up schedule due to geographic distance from the Siteman Cancer Center should not knowingly be registered.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-09-29 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety of the vaccine regimen as measured by grade and frequency of adverse events | 1 year
  -Toxicity will be characterized according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 (CTCAE). -Subjects who are immunized with the synthetic long peptide vaccine will be evaluated at the time of each vaccination. Follow-up on subject well-being will be performed by telephone on the first or second day after each vaccination.

SECONDARY OUTCOMES:
Immunogenicity of the vaccine regimen as measured by ELISPOT analyses | 1 year
  * ELISPOT analyses is a surrogate for CD8 T cell function
  * The quantity and quality of antigen-specific CD8 T cells is determined
  * The ELISPOT analysis is based on measuring the frequencies of IFN-γ producing T cells in response to polyepitope antigen
Immunogenicity of the vaccine regimen as measured by multiparametric flow cytometry | 1 year
  * Multiparametric flow cytometry is a surrogate for CD8 T cell function
  * The quantity and quality of antigen-specific CD8 T cells is determined
  * Multiparametric flow cytometry assesses phenotypic as well as functional characteristics of epitope-specific CD8 T cells

CONTACTS AND LOCATIONS:
Overall Officials: Williams E Gillanders, M.D., Principal Investigator — Washington University School of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu